CLINICAL TRIAL: NCT00066846
Title: A Multicenter Study of the Anti-VEGF Monoclonal Antibody Bevacizumab (Avastin®) Plus 5-Fluorouracil/Leucovorin in Patients With Metastatic Colorectal Cancers That Have Progressed After Standard Chemotherapy
Brief Title: Bevacizumab Plus Fluorouracil and Leucovorin in Treating Patients With Locally Advanced or Metastatic Stage IV Colorectal Cancer That Has Progressed After Standard Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000320506; CTEP-TRC-0301
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV rectal cancer; recurrent rectal cancer; stage IV colon cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin

INTERVENTIONS:
Biological: bevacizumab
Drug: fluorouracil
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Bevacizumab may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy such as fluorouracil and leucovorin use different ways to stop tumor cells from dividing so they stop growing or die. Combining bevacizumab with fluorouracil and leucovorin may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining bevacizumab with fluorouracil and leucovorin in treating patients who have locally advanced or metastatic stage IV colorectal cancer that has progressed after standard chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients treated with bevacizumab, fluorouracil, and leucovorin calcium for stage IV colorectal cancer that has progressed after standard chemotherapy.
* Determine the time to progression and overall survival of patients treated with this regimen.
* Determine the safety of administering "bolus" and continuous infusion fluorouracil and leucovorin calcium in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study. Patients receive 1 of 2 treatment regimens.

* Regimen I: Patients receive bevacizumab IV on days 1, 15, 29, and 42 (every 2 weeks) and leucovorin calcium (CF) IV over 2 hours and fluorouracil (5-FU) IV bolus on days 1, 8, 15, 22, 29, and 36.
* Regimen II: Patients receive bevacizumab as in regimen I and CF IV over 2 hours and 5-FU IV bolus followed by a continuous infusion over 22 hours on days 1, 2, 15, 16, 29, 30, 43, and 44.

For both regimens, courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for tumor response and survival.

PROJECTED ACCRUAL: Various NCI-designated Clinical Cancer Centers and other medical institutions across the United States will participate in this study. A total of 35-125 patients will be accrued for this study within 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal adenocarcinoma

  * Stage IV (metastatic) disease
  * Not curable by surgery or radiotherapy
* Must have received prior standard chemotherapy regimens, including oxaliplatin and irinotecan, and meet both of the following criteria:

  * Disease progression during or after irinotecan-based chemotherapy for metastatic disease OR relapsed disease within 6 months after adjuvant irinotecan-based therapy
  * Disease progression during or after oxaliplatin-based chemotherapy for metastatic disease OR relapsed disease within 6 months after adjuvant oxaliplatin-based therapy
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)
* No evidence of bleeding diathesis or coagulopathy

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST less than 5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 5 times ULN
* PT and INR no greater than 1.5 times ULN
* PTT no greater than ULN

Renal

* Creatinine no greater than 1.5 times ULN
* Proteinuria less than grade 1 OR
* Proteinuria less than 500 mg/24 hours

Cardiovascular

* No prior stroke
* No uncontrolled high blood pressure
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart disease
* No thromboembolism within the past 6 months

Other

* Chemonaive
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* No significant traumatic injury within the past 6 weeks
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to bevacizumab or other study agents
* No active infection
* No psychiatric illness or social situation that would preclude study compliance
* No serious nonhealing wound (including wounds healing by secondary intention), ulcer, or bone fracture
* No CNS disease, including either of the following:

  * Primary brain tumor
  * Seizures not controlled with standard medical therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 8 weeks since prior monoclonal antibody therapy
* No prior bevacizumab

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior major radiotherapy (e.g., chest or bone palliative radiotherapy)

Surgery

* More than 6 weeks since prior major surgical procedure or open biopsy
* More than 7 days since prior fine needle aspiration or core biopsy
* No concurrent surgery

Other

* Recovered from prior therapy
* At least 3 weeks since prior cytotoxic agents
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation of venous access devices allowed provided PT/INR or PTT criteria are met
* No concurrent chronic aspirin (greater than 325 mg/day) or nonsteroidal anti-inflammatory drugs
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen X. Chen, MD, Principal Investigator — NCI - Investigational Drug Branch
Locations (33):
- United States (33):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Cancer Care of Maine, Bangor, Maine
  - Saint Joseph Mercy Health System, Ann Arbor, Michigan
  - St. Mary's/Duluth Clinic Cancer Center, Duluth, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Sioux Valley Clinics - Oncology, Sioux Falls, South Dakota
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Result] Chen HX, Mooney M, Boron M, Vena D, Mosby K, Grochow L, Jaffe C, Rubinstein L, Zwiebel J, Kaplan RS. Phase II multicenter trial of bevacizumab plus fluorouracil and leucovorin in patients with advanced refractory colorectal cancer: an NCI Treatment Referral Center Trial TRC-0301. J Clin Oncol. 2006 Jul 20;24(21):3354-60. doi: 10.1200/JCO.2005.05.1573. PMID 16849749